CLINICAL TRIAL: NCT01593748
Title: A Randomized, Open-label, Phase II, Multi-center Trial of Gemcitabine (G) With Pazopanib (P) or Gemcitabine (G) With Docetaxel (T) in Previously Treated Subjects With Advanced Soft Tissue Sarcoma
Brief Title: A Phase II Trial Comparing Gemcitabine and Pazopanib Versus Gemcitabine and Docetaxel for Patients With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101644; PAZ115785 (Other: GlaxoSmithKline); CPZP034BUS1T (Other: Novartis)
Record Dates: First submitted 2012-05-04; First posted 2012-05-08 (Estimated); Results first posted 2020-04-06 (Actual); Last update posted 2020-04-06 (Actual); Status verified 2020-03

CONDITIONS: Sarcoma
Keywords: Sarcoma; Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Gemcitabine; pazopanib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Patients in Group 1 will get Gemcitabine 1000 mg/m2 intravenously on Day 1 and Day 8 and Pazopanib 800mg by mouth daily on a 21 day cycle. Cycles will continue until disease progression or patient withdrawal.
  Interventions: Drug: Gemcitabine and Pazopanib
- Standard of Care (Active Comparator): Patients in Group 2 will get Gemcitabine 900 mg/m2 intravenously on Day 1 and Day 8. Additionally on Day 8, patients will have Docetaxel 100 mg/m2 given intravenously. on a 21 day cycle. If disease progression occurs on this treatment, patients will have the option to receive treatment with Gemcitabine and Pazopanib (group 1).
  Interventions: Drug: Gemcitabine and Docetaxel

INTERVENTIONS:
Drug: Gemcitabine and Pazopanib — Gemcitabine 1000 mg/m2 by IV on day 1 and day 8 of a 21 day cycle. Pazopanib 800 mg by oral tablet daily for a 21 day cycle.
  Arms: Experimental
Drug: Gemcitabine and Docetaxel — Gemcitabine 900 mg/m2 by IV on day 1 and day 8 of a 21 day cycle. Docetaxel 100 mg/m2 by IV on day 8 of a 21 day cycle.
  Arms: Standard of Care

SUMMARY:
This study is for adult subjects with advanced tissue sarcoma. The study involves the drugs Pazopanib (Votrient), Gemcitabine (Gemzar), and Docetaxel (Taxotere). The purpose of this study is to test the effectiveness and safety of Gemcitabine and Pazopanib compared with Gemcitabine and Docetaxel in participants with soft tissue sarcoma.

DETAILED DESCRIPTION:
The purpose of this study is to test the effectiveness and safety of Gemcitabine and Pazopanib compared with Gemcitabine and Docetaxel in participants with soft tissue sarcoma. Screening tests will be done to ensure subjects are eligible to participate in this study. If the exams, tests and procedures show that subjects can be in the study, and they choose to take part, then they will be "randomized" into one of the two study groups: Group 1 or Group 2. Subjects in Group 1 will receive Gemcitabine 1000 mg/m2 intravenously (directly into a vein) on Day 1 and Day 8 and Pazopanib 800mg by mouth daily. Subjects in Group 2 will receive Gemcitabine 900 mg/m2 intravenously on Day 1 and Day 8 and Docetaxel 100 mg/m2 intravenously on Day 8. Both groups will be in 21 day cycles. Both groups will be asked to complete "quality of life" questionnaires, on their first visit, then at 6 weeks (2nd cycle), 18 weeks (6th cycle) and at the end of study treatment. Subjects will be followed for up to 2 years.

ELIGIBILITY:
* Subjects must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
* Age ≥ 18 years or legal age of consent if greater than 18 years.
* Histologically or cytologically confirmed diagnosis of sarcoma of soft tissue. (Patients with liposarcoma, bone sarcoma or GIST will be excluded).
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Subjects must have metastatic and/or locally advanced or locally recurrent disease that is not amenable to curative surgical resection.
* A minimum of 1 and a maximum of 3 prior chemotherapy regimens for recurrent/metastatic disease. Patients eligible for an anthracycline should have received a prior anthracycline containing regimen. Patients who decline or are not eligible for anthracycline treatment may be considered for this protocol as a first line treatment.
* Patients must have measurable disease by RECIST 1.1. or cutaneous disease amenable to serial measurements should be present. Measurable disease (a 'target' lesion) is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be ≥ 10 mm when measured by CT (CT scan slice thickness no greater than 5 mm); ≥ 10 mm caliper measurement by clinical exam (lesions which cannot be accurately measured with calipers should be recorded as non-measurable); and ≥ 20 mm by chest x-ray.
* Able to swallow and retain oral medication.
* Adequate organ system function
* A female is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal

Subjects not using hormone replacement therapy (HRT) must have experienced total cessation of menses for ≥ 1 year and be greater than 45 years in age, OR, in questionable cases, have a follicle stimulating hormone (FSH) value > 40 mIU/mL and an estradiol value < 40pg/mL (< 140 pmol/L).

Subjects using HRT must have experienced total cessation of menses for >= 1 year and be greater than 45 years of age OR have had documented evidence of menopause based on FSH and estradiol concentrations prior to initiation of HRT.

-- Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. Acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:

* Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product
* Oral contraceptive, either combined or progestogen alone
* Injectable progestogen
* Implants of levonorgestrel
* Estrogenic vaginal ring
* Percutaneous contraceptive patches
* Intrauterine device (IUD) or intrauterine system (IUS) with a documented failure rate of less than 1% per year
* Male partner sterilization (vasectomy with documentation of azoospermia) prior to the female subject's entry into the study, and this male is the sole partner for that subject
* Double barrier method: condom and an occlusive cap (diaphragm or cervical/vault caps) with a vaginal spermicidal agent (foam/gel/film/cream/suppository)

Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.

Exclusion Criteria

* Prior therapy with pazopanib, gemcitabine or docetaxel.
* Any concern for hypersensitivity to pazopanib, gemcitabine or docetaxel.
* Prior malignancy. Note: Subjects who have had another malignancy and have been disease-free for 3 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.
* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

  * Active peptic ulcer disease
  * Known intraluminal metastatic lesion/s with risk of bleeding
  * Inflammatory bowel disease (e.g. ulcerative colitis, Crohn's disease), or other gastrointestinal conditions with increased risk of perforation
  * History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.

Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

* Malabsorption syndrome
* Major resection of the stomach or small bowel and experiencing the "dumping" syndrome.

  * Presence of uncontrolled infection.
  * Prior mediastinal radiation
  * Corrected QT interval (QTc) > 480 msecs using Bazett's formula.
  * History of any one or more of the following conditions within the past 6 months:
* Cardiac angioplasty or stenting
* Myocardial infarction
* Unstable angina
* Coronary artery bypass graft surgery
* Symptomatic peripheral vascular disease
* Pneumonitis

  * Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA) (Appendix D).
  * Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥ 150 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].

Note: Initiation or adjustment of antihypertensive medication(s) is permitted prior to study entry. BP must be re-assessed on two occasions that are separated by a minimum of 1 hour; on each of these occasions, the mean (of 3 readings) SBP/DBP values from each BP assessment must be < 150/90 mmHg in order for a subject to be eligible for the study.

-History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks prior to registration and are fully anti-coagulated are eligible.

* Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
* Evidence of active bleeding or bleeding diathesis.
* Known endobronchial lesions and/or lesions infiltrating major pulmonary Hemoptysis in excess of 2.5 mL (or one half teaspoon) within 8 weeks of first dose of study drug.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
* Unable or unwilling to discontinue use of prohibited medications listed in Section 5.2.3 for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
* Treatment with any of the following anti-cancer or non-oncologic investigational therapies:

  * radiation therapy, surgery or tumor embolization within 14 days prior to registration.
  * chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or 2.5 half-lives of a drug (whichever is longer) prior to registration.
  * non-oncologic investigational products within 30 days or 5 halflives, whichever is longer.
* Any ongoing toxicity from prior anti-cancer therapy that is >Grade 1 and/or that is progressing in severity, except alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Y. Reuben, MD, Principal Investigator — Medical University of South Carolina Hollings Cancer Center
Locations (8):
- United States (8):
  - The University of Arizona Cancer Center, Tucson, Arizona
  - University of Colorado Cancer Center, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Washington University at St. Louis, St Louis, Missouri
  - University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Xin G, Wang M, Jiao LL, Xu GB, Wang HY. Protein-to-creatinine ratio in spot urine samples as a predictor of quantitation of proteinuria. Clin Chim Acta. 2004 Dec;350(1-2):35-9. doi: 10.1016/j.cccn.2004.06.019. PMID 15530457
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: Patients in Group 1 will get Gemcitabine 1000 mg/m2 intravenously on Day 1 and Day 8 and Pazopanib 800mg by mouth daily on a 21 day cycle. Cycles will continue until disease progression or patient withdrawal.
  Gemcitabine and Pazopanib: Gemcitabine 1000 mg/m2 by IV on day 1 and day 8 of a 21 day cycle.
  Pazopanib 800 mg by oral tablet daily for a 21 day cycle.
- Standard of Care: Patients in Group 2 will get Gemcitabine 900 mg/m2 intravenously on Day 1 and Day 8. Additionally on Day 8, patients will have Docetaxel 100 mg/m2 given intravenously. on a 21 day cycle. If disease progression occurs on this treatment, patients will have the option to receive treatment with Gemcitabine and Pazopanib (group 1).
  Gemcitabine and Docetaxel: Gemcitabine 900 mg/m2 by IV on day 1 and day 8 of a 21 day cycle.
  Docetaxel 100 mg/m2 by IV on day 8 of a 21 day cycle.
Period: Overall Study
Arm/Group | Experimental | Standard of Care
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental | Standard of Care | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.93 (13.76) | 54.6 (14.10) | 56.27 (13.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 22 | 46
  Male | 21 | 23 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 37 | 43 | 80
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 8 | 11
  White | 36 | 33 | 69
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Months of Progression-free Survival
Description: To estimate the PFS of the combination of G+P or G+T in patients with metastatic and/or locally advanced or recurrent STS. Progression free survival is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
Time Frame: minimum of 18 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Experimental | Standard of Care
Number analyzed (Participants) | 45 | 45
months | 4.1 [2.4 to 8.6] | 4.1 [2.7 to 11.4]

2. Primary Outcome: Rate of Participants With Grade 3 or Higher Toxicity
Description: Toxicity is graded according to the CTCAE v 4.
Time Frame: 30 days post end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Standard of Care
Number analyzed (Participants) | 45 | 45
Participants | 39 | 39

3. Secondary Outcome: Hazard Ratio
Description: Hazard ratio is defined as the rate of survival in the experimental group versus the standard of care group. A hazard ratio of greater than one or less than one means that survival was better in one of the groups.
Time Frame: minimum of 18 months
Measure: Number (95% Confidence Interval); unit: hazard ratio
Arm/Group | Experimental | Standard of Care
Number analyzed (Participants) | 45 | 45
hazard ratio | 1.2 [0.7 to 2.0] | NA [NA to NA] — Not applicable; outcome is expressed as a single ratio

4. Secondary Outcome: Average Score of Quality of Life
Description: To estimate the quality of life of patient with metastatic an/or locally advanced recurrent STS using the Quality of Life Questionnaire (QLQ-C30). The QLQ-C30 is scored on a scale from 0-100 with "0" indicating "never" and "100" indicating "always" in regard the the participants' experience of fatigue, nausea/vomiting, pain, disponae, insomnia, appetite loss, constipation, diarrhea, financial concerns at 4 time points through the study.
Time Frame: Baseline, Cycle 2, Cycle 6 and End of Treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental | Standard of Care
Number analyzed (Participants) | 45 | 45
score on a scale
  Fatigue at baseline | 61.79 (27.89) | 67.12 (23.44)
  Nausea/Vommiting at baseline | 91.06 (14.48) | 90.99 (16.94)
  Pain at baseline | 61.38 (32.80) | 74.77 (25.65)
  Dysponae at baseline | 22.76 (32.86) | 21.62 (29.62)
  Insomnia at baseline | 45.53 (39.97) | 36.04 (30.81)
  Appetite loss at baseline | 22.76 (32.01) | 15.32 (26.75)
  Constipation at baseline | 14.63 (26.92) | 15.32 (23.03)
  Diarrhea at baseline | 4.88 (11.93) | 8.11 (16.49)
  Financial at baseline | 37.40 (40.96) | 32.43 (34.68)
  Fatigue at cycle 2 | 52.89 (23.85) | 55.09 (25.06)
  Nausea/Vomitting at cycle 2 | 80.67 (17.13) | 93.75 (9.60)
  Pain at cycle 2 | 66.00 (26.56) | 83.33 (20.85)
  Dyspnoae at cycle 2 | 24.00 (24.57) | 26.39 (24.04)
  Insomnia at cycle 2 | 42.67 (34.05) | 38.89 (28.94)
  Appetite loss at cycle 2 | 36.11 (32.48) | 26.39 (32.57)
  Constipation at cycle 2 | 13.33 (21.52) | 23.61 (25.02)
  Diarrhea at cycle 2 | 4.88 (11.93) | 8.11 (16.49)
  Financial at cycle 2 | 26.67 (34.69) | 22.22 (27.22)
  Fatigue at cycle 6 | 64.44 (11.48) | 51.11 (30.63)
  Nausea/vommiting at cycle 6 | 86.67 (7.03) | 8.05 (95.00)
  Pain at cycle 6 | 80.00 (23.31) | 78.33 (30.48)
  Dyspnoae at cycle 6 | 10.00 (16.10) | 43.33 (22.50)
  Insomnia at cycle 6 | 23.33 (16.10) | 33.33 (27.22)
  Appetite loss at cycle 6 | 26.67 (34.43) | 30.00 (24.60)
  Constipation at cycle 6 | 13.33 (17.21) | 13.33 (23.31)
  Diarrhea at cycle 6 | 36.67 (24.60) | 20.00 (23.31)
  Financial at cycle 6 | 23.33 (31.62) | 20.00 (23.31)
  Fatigue at end of study | 49.81 (22.74) | 49.77 (25.77)
  Nausea/vomitting at end of study | 75.86 (23.82) | 92.36 (12.02)
  Pain at end of study | 53.45 (32.85) | 72.92 (24.48)
  Dysponae at end of study | 31.03 (33.25) | 34.72 (28.62)
  Insomnia at end of study | 48.28 (36.28) | 37.50 (26.58)
  Appetite loss at end of study | 37.93 (33.00) | 23.61 (28.62)
  Constipation at end of study | 17.24 (24.59) | 29.17 (30.00)
  Diarrhea at end of study | 21.43 (22.62) | 15.28 (24.04)
  Financial at end of study | 39.60 (39.29) | 29.17 (33.06)

5. Secondary Outcome: Response Rate
Description: Response rate is defined as follows:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study
Time Frame: minimum of 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental | Standard of Care
Number analyzed (Participants) | 43 | 45
Participants
  Complete Response | 0 | 0
  Partial Response | 5 | 8
  Stable Disease | 24 | 21
  Progressive Disease | 14 | 16

ADVERSE EVENTS:
Time Frame: study enrollment to 30 days from last treatment; inclusive of crossover treatment
Description: AE data was collected from subjects at every clinic visit and day 1 of every cycle.
Arm/Group | Experimental | Standard of Care
All-Cause Mortality (participants affected / at risk) | 32/45 | 30/45
Serious Adverse Events (participants affected / at risk) | 28/45 | 31/45
Other Adverse Events (participants affected / at risk) | 45/45 | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=45) | Standard of Care (N=45)
Fever (General disorders) | 3 | 3
Nausea (Gastrointestinal disorders) | 2 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Asystole (Cardiac disorders) | 1 | 0
Atrial Fibrilation (Cardiac disorders) | 1 | 1
Heart Failure (Cardiac disorders) | 1 | 0
Pericardial Tamponade (Cardiac disorders) | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1
Pain (General disorders) | 1 | 1
Edema Limbs (General disorders) | 0 | 2
Edema Trunk (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 2
Bacterial Infection (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Spinal Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Platelet Count Decrease (Investigations) | 2 | 2
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Bleeding from Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischemia Cerebrovascular (Nervous system disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone Pain/Right leg (Musculoskeletal and connective tissue disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Acute Left Lung Pneumonia/Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thromboembolic Event (Vascular disorders) | 1 | 0
Other Infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=45) | Standard of Care (N=45)
Fatigue (General disorders) | 34 | 28
Platelet Count Decreased (Investigations) | 34 | 33
Nausea (Gastrointestinal disorders) | 31 | 18
Anemia (Blood and lymphatic system disorders) | 27 | 32
Constipation (Gastrointestinal disorders) | 13 | 19
Neutrophil Count Decreased (Investigations) | 26 | 11
Edema Limbs (General disorders) | 7 | 16
Vomiting (Gastrointestinal disorders) | 25 | 5
Pain (General disorders) | 16 | 16
Diarrhea (Gastrointestinal disorders) | 22 | 14
Alanine Aminotransferase Increased (Investigations) | 20 | 12
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 14
Anorexia (Metabolism and nutrition disorders) | 16 | 13
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 13
White Blood Cell Decreased (Investigations) | 19 | 13
Aspartate Aminotransferase Increased (Investigations) | 20 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Dysgeusia (Nervous system disorders) | 5 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 12
Fever (General disorders) | 8 | 11
Hypokalemia (Metabolism and nutrition disorders) | 7 | 11
Mucositis Oral (Gastrointestinal disorders) | 7 | 11
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 11
Alkaline Phosphatase Increased (Investigations) | 13 | 10
Headache (Nervous system disorders) | 15 | 10
Lymphocyte Count Decreased (Investigations) | 9 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 9
Hyponatremia (Metabolism and nutrition disorders) | 6 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 7
Insomnia (Psychiatric disorders) | 9 | 7
Dizziness (Nervous system disorders) | 7 | 6
Nail Discoloration (Skin and subcutaneous tissue disorders) | 0 | 6
Abdominal Pain (Gastrointestinal disorders) | 7 | 5
Creatinine Increased (Investigations) | 2 | 5
Depression (Psychiatric disorders) | 0 | 5
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 5
Hypernatremia (Metabolism and nutrition disorders) | 3 | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 5
Palmarplantar Erythrodysesthesia Syndrome (Skin and subcutaneous tissue disorders) | 5 | 5
Hypertension (Vascular disorders) | 16 | 3
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Blood Bilirubin Increased (Investigations) | 6 | 2
Noncardiac Chest Pain (General disorders) | 5 | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 5 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT01593748/Prot_SAP_000.pdf